CLINICAL TRIAL: NCT05637021
Title: Study on the Influencing Factors of Intestinal Microecology Changes Before and After Colonoscopy
Brief Title: Effect of Carbon Dioxide Insufflation and Appendix on the Restoration of Intestinal Microecology After Colonoscopy.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-014
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Colonoscopy; Gastrointestinal Microbiome; Appendix; Carbon Dioxide Insufflation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — feces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Healthy people were randomly divided into CO2 group and control group, with 20 cases in each group. After bowel preparation, volunteers underwent colonoscopy, with air routinely insufflated into the control group during colonoscopy.
- Carbon dioxide group: Healthy people were randomly divided into CO2 group and control group, with 20 cases in each group. After bowel preparation, volunteers underwent colonoscopy, with CO2 insufflated into the control group during colonoscopy.
  Interventions: Other: Carbon dioxide insufflated during colonoscopy
- After appendectomy group: Volunteers after appendectomy were included in the appendectomy group. After bowel preparation, all volunteers underwent colonoscopy, air routinely insufflated into the appendectomy group.

INTERVENTIONS:
Other: Carbon dioxide insufflated during colonoscopy — Carbon dioxide is insufflated to dilate the bowel lumen during colonoscopy.Record the amount of gas insufflated during colonoscopy.
  Groups: Carbon dioxide group

SUMMARY:
The goal of this observational study is to learn about Influencing factors of intestinal microecological changes before and after colonoscopy. The main questions it aims to answer are:

* [question 1] The process of colonoscopic gas insufflation affects the intestinal microecology. Will the use of carbon dioxide gas insufflation can reduce the changes of intestinal microecology after colonoscopy?
* [question 2] Can the appendix act as a reservoir for microorganisms to accelerate the recovery of intestinal microecology after colonoscopy？

Participants will be asked to accept colonoscopy for once. Group 1(Control group) will be insufflated air during the colonoscopy; Group 2(Carbon dioxide group) will be insufflated carbon dioxide during the colonoscopy; Group 3(After appendectomy group) will be insufflated air during the colonoscopy.

Since Group 1 is comparison group, the investigators will compare Group 2 to see if carbon dioxide gas insufflation can reduce the changes of intestinal microecology after colonoscopy. Meanwhile, compare Group 3 to see if the appendix can accelerate the recovery of intestinal microecology after colonoscopy.

DETAILED DESCRIPTION:
Usually, gastroenteroscopy requires gas insufflation to expand the lumen to facilitate endoscopic insertion and detailed observation of the mucosa. In the past, the use of air as an insufflation gas in endoscopic operations was simple and inexpensive, but because its main component was nitrogen, it was difficult to be absorbed by the gastrointestinal mucosa. Therefore, the endoscopist often needs to fully aspirate the gas when the procedure is completed. However, studies have shown that about 50% of patients still complain of abdominal pain after colonoscopy, and 12% of patients still have severe abdominal pain even after 24 hours. In contrast, carbon dioxide (CO2) has been used in endoscopy of the digestive tract in recent years because it can be rapidly absorbed by the gastrointestinal mucosa, and has attracted the attention of endoscopists.

The gastrointestinal mucosa absorbs CO2 at a rate 160 times faster than nitrogen. Because of this property, many people consider replacing air in endoscopic operations. Its potential value was first demonstrated in animal tests: the recovery time of intestinal lumen dilation and increased intraluminal pressure was significantly shortened after intestinal lumen injection of CO2 in rats. Meta-analysis showed no significant difference in safety, gas volume, or cecal intubation rate between the two groups for CO2 insufflation during colonoscopy, but less postoperative abdominal pain, abdominal distention, and less postoperative gastrointestinal exhaust in the CO2 group. The low postoperative pain score and low increase in abdominal circumference may be due to the rapid absorption of CO2 by the gastrointestinal mucosa, suggesting that residual gas after colonoscopy is the main cause of abdominal pain. CO2 is a non-flammable gas that is safe for electroresection and has been widely used in laparoscopic surgery. For patients with chronic obstructive pulmonary disease (COPD) who require endoscopy, it is worth exploring whether the use of CO2 in endoscopy causes CO2 retention. In one study of 77 endoscopic participants with obstructive ventilation dysfunction and 308 endoscopic participants without concomitant obstructive ventilation dysfunction, there was no difference in end-tidal volume CO2 between the two groups, and the peak tidal volume CO2 peak was less than 60 mmHg in both groups, suggesting that endoscopic use of CO2 is still safe for people with concomitant obstructive ventilation dysfunction.

The current study has found that the intestinal preparation of the colonoscopy, as well as the colonoscopy operation itself, has a certain impact on the intestinal microbiome, although this effect can be partially recovered over a period of time, but the current study has found that this change may also be permanent, but whether it will cause long-term metabolic, immune or clinical changes in the host is unknown. Compared with conventional air injection, CO2 may change less about the hypoxic environment of the intestine, thereby reducing the impact on the normal intestinal microbiome.

Based on this hypothesis, the investigators will conduct randomized, controlled experiments to investigate the effects of conventional air and CO2 insufflation on the intestinal microbiome and metabolites.

In addition, some studies have called the appendix a "reservoir" of gut microbes. First, the mucosal flora of the appendix is similar to the rest of the colon; Secondly, the fecal microbiota composition of mice changed after appendectomy. The appendix preserves a small amount of intestinal bacteria as "seeds", once the intestinal flora is imbalanced, the "seed bank" will be used for cultivation, when the appendix is removed, it is equivalent to the "seed bank" is destroyed, so once the intestinal flora is imbalanced, there may be a delay in the recovery of the intestinal microecology.

Based on this hypothesis, the investigators will conduct controlled experiments to compare the intestinal microbiome recovery after colonoscopy in healthy people and people after appendectomy, and explore the impact of appendix on intestinal microbiome recovery.

This study was a single-center study, and 20 cases were initially included in the control group, CO2 group and after appendectomy group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years old, gender is not limited, no underlying diseases;
* BMI between 18.5-23.9 kg/m2;
* Fecal Bristol score type III-IV in the past week;
* No history of alcohol consumption or alcohol consumption equivalent to ethanol should not exceed 140g per week for men and 70g per week for women.
* Add a criterion to after appendectomy group:Patients who underwent appendectomy in the Department of General Surgery of Zhongshan Hospital Xiamen University within 3 years.

Exclusion Criteria:

* Those who use antibiotics, antifungal drugs, antiviral drugs, probiotics, prebiotics, synbiotics and drugs that may affect the intestinal microecology within 1 month;
* Those who have acute enteritis or chronic enteritis and other diagnosed chronic bowel diseases in the past 1 month;
* Those who have digestive symptoms such as blood in the stool, constipation, bloating, abdominal pain, diarrhea and so on in the past 1 month
* History of digestive surgery (including gastrointestinal polyp resection, gastrointestinal tumor surgery and diversion surgery, etc.).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The patients in the after appendectomy group were patients who underwent appendectomy in the Department of General Surgery, Zhongshan Hospital Xiamen University within 3 years.
  The other volunteers are residents of Xiamen City.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The intestinal microbiota composition | Before bowel cleansing, after colonoscopy, 7、14 and 28 days after the treatment
  Changes in the intestinal microbiome are observed by detecting the feces at the specific time point.Then, factors affecting the recovery of the intestinal microbiome are assessed based on their changes.

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhi Xu, Principal Investigator — Zhongshan Hospital Xiamen University
Locations (1):
- Zhongshan Hospital Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication.
Access Criteria: To the public.

REFERENCES:
- [Background] Wu J, Hu B. The role of carbon dioxide insufflation in colonoscopy: a systematic review and meta-analysis. Endoscopy. 2012 Feb;44(2):128-36. doi: 10.1055/s-0031-1291487. Epub 2012 Jan 23. PMID 22271023
- [Background] Eckburg PB, Bik EM, Bernstein CN, Purdom E, Dethlefsen L, Sargent M, Gill SR, Nelson KE, Relman DA. Diversity of the human intestinal microbial flora. Science. 2005 Jun 10;308(5728):1635-8. doi: 10.1126/science.1110591. Epub 2005 Apr 14. PMID 15831718
- [Background] Masahata K, Umemoto E, Kayama H, Kotani M, Nakamura S, Kurakawa T, Kikuta J, Gotoh K, Motooka D, Sato S, Higuchi T, Baba Y, Kurosaki T, Kinoshita M, Shimada Y, Kimura T, Okumura R, Takeda A, Tajima M, Yoshie O, Fukuzawa M, Kiyono H, Fagarasan S, Iida T, Ishii M, Takeda K. Generation of colonic IgA-secreting cells in the caecal patch. Nat Commun. 2014 Apr 10;5:3704. doi: 10.1038/ncomms4704. PMID 24718324
- [Result] Jalanka J, Salonen A, Salojarvi J, Ritari J, Immonen O, Marciani L, Gowland P, Hoad C, Garsed K, Lam C, Palva A, Spiller RC, de Vos WM. Effects of bowel cleansing on the intestinal microbiota. Gut. 2015 Oct;64(10):1562-8. doi: 10.1136/gutjnl-2014-307240. Epub 2014 Dec 19. PMID 25527456
- [Result] Drago L, Toscano M, De Grandi R, Casini V, Pace F. Persisting changes of intestinal microbiota after bowel lavage and colonoscopy. Eur J Gastroenterol Hepatol. 2016 May;28(5):532-7. doi: 10.1097/MEG.0000000000000581. PMID 27015015
- [Result] Nagata N, Tohya M, Fukuda S, Suda W, Nishijima S, Takeuchi F, Ohsugi M, Tsujimoto T, Nakamura T, Shimomura A, Yanagisawa N, Hisada Y, Watanabe K, Imbe K, Akiyama J, Mizokami M, Miyoshi-Akiyama T, Uemura N, Hattori M. Effects of bowel preparation on the human gut microbiome and metabolome. Sci Rep. 2019 Mar 11;9(1):4042. doi: 10.1038/s41598-019-40182-9. PMID 30858400